CLINICAL TRIAL: NCT01537419
Title: Attachment Based Family Therapy (ABFT) for Suicidal Adolescents
Brief Title: Attachment Based Family Therapy for Suicidal Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1304001985; R01MH091059-01A1 (NIH)
Record Dates: First submitted 2012-02-13; First posted 2012-02-23 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Suicide; Depression; Family Relationships
Keywords: Suicide; Depression; Family Relationships
MeSH Terms: conditions — Suicide; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family-Enhanced Non-directive Supportive Therapy (Active Comparator): Family-Enhanced Non-directive Supportive Therapy (FE-NST) is a 16 week therapy designed to control for the non-specific effects of psychotherapy with suicidal youth. FE-NST aims toward relief or reduction of symptoms without expectation of change in the basic personality structure. We have added a parent component to: a) control for parent involvement and b) improve the generalizability and safety of the FE-NST treatment. This enhancement consists of 5 potential parent sessions beginning with a family safety plan in the initial treatment session that will be monitored regularly throughout the treatment. The remaining 4 parent psycho-education sessions offer parents knowledge, skills and support to improve management of the suicidal teen.
  Interventions: Behavioral: Family-Enhanced Non-directive Supportive Therapy
- Attachment-Based Family Therapy (Experimental): Although ABFT therapists implement behavior focused and psychoeducational interventions, the model is primarily a process oriented, emotion focused treatment guided by a semi-structured treatment protocol. ABFT aims to improve the family's capacity for problem solving, affect regulation, and organization. This strengthens family cohesion which can buffer against depression, suicidal thinking, and risk behaviors.
  Interventions: Behavioral: Attachment-Based Family Therapy

INTERVENTIONS:
Behavioral: Attachment-Based Family Therapy — Although ABFT therapists implement behavior focused and psychoeducational interventions, the model is primarily a process oriented, emotion focused treatment guided by a semi-structured treatment protocol. ABFT aims to improve the family's capacity for problem solving, affect regulation, and organization. This strengthens family cohesion which can buffer against depression, suicidal thinking, and risk behaviors.
  Arms: Attachment-Based Family Therapy
Behavioral: Family-Enhanced Non-directive Supportive Therapy — Family-Enhanced Non-directive Supportive Therapy (FE-NST) is a 16 week therapy designed to control for the non-specific effects of psychotherapy with suicidal youth. FE-NST aims toward relief or reduction of symptoms without expectation of change in the basic personality structure. We have added a parent component to: a) control for parent involvement and b) improve the generalizability and safety of the FE-NST treatment. This enhancement consists of 5 potential parent sessions beginning with a family safety plan in the initial treatment session that will be monitored regularly throughout the treatment. The remaining 4 parent psycho-education sessions offer parents knowledge, skills and support to improve management of the suicidal teen.
  Arms: Family-Enhanced Non-directive Supportive Therapy

SUMMARY:
This study will evaluate the efficacy of attachment based family therapy (ABFT) for treatment of suicidality in adolescents. The study will compare 16 weeks of treatment with ABFT to a control condition Family Enhanced Non-directive Supportive Therapy (FE-NST).

DETAILED DESCRIPTION:
Suicide is the third leading cause of death for American adolescents. Nearly one million adolescents a year attempt suicide and about 500,000 adolescents a year are admitted to psychiatric hospitals for suicide attempts or serious suicidal ideation. This leads to high emotional costs for families and financial cost for the health system. Yet, no medication, and less than 10 psychotherapy studies have focused on suicidal youth and findings are mixed. There has been a call for new and innovative approaches for depression treatment highlights the need for alternative interventions for suicidal youth as well. Attachment-Based Family Therapy (ABFT) offers a promising alternative to prior treatments. It is a manualized family therapy targeting processes associated with suicide and depression. ABFT seeks to improve the adolescent-caregiver relationship by increasing the family's capacity for discussing and negotiating affectively charged issues in the relationship. Improvements in the attachment relationship provide adolescents with improved capacity for affect regulation and the ability to use the caregiver as a source of protection and support. These strengths buffer adolescents against suicide and other risk behaviors. Four studies have demonstrated that ABFT can reduce suicidal ideation and depressive symptoms with an average effect size of .97. Unfortunately, interpretation of these studies is compromised by lack of a controlled comparison treatment. This study aims to test the efficacy of ABFT using a comparison group that controls for treatment dose, duration, therapist expertise, ecological factors, and family involvement. The study includes one year follow-up data, assessment staff blind to treatment condition and tests of the purported active ingredients of ABFT. Putative change processes will be tested including: a)adolescents' expectancies for parent availability, b) emotion regulation during parent-adolescent conflict discussions, and c) resolution of loss and abuse. To test this, Dr. Kobak, a leading adolescent attachment researcher, will use the Adult Attachment Interview and observational coding of the family interaction task to test these treatment mechanisms. If successful, the findings will provide evidence for both the efficacy and specificity of a family based treatment mechanism. The investigators will recruit and randomize 130 adolescents to 16 weeks of ABFT or Family-Enhanced Non-directive Supportive Therapy (FE-NST). Assessments will be conducted at baseline, 8, 16, 32 and 52 weeks. The primary and secondary aims assess whether ABFT reduces suicidal ideation, depression, family conflict, and future suicide attempts more effectively than control. Exploratory aims test a) whether ABFT can improve parent adolescent attachment, b) if attachment mediates outcome, and if a history of trauma, parental depression or family conflict moderate outcome. The study targets adolescents with severe and persistent suicidal ideation selected from inner city, minority youth.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 12 and 18
* Adolescents endorse severe suicidal ideation (SIQ-JR > 31) and moderate depression (BDI-II > 20) at two time points (1 to 3 days)
* At least one primary parent or caregiver must participate in the assessment and treatment. This could be a biological parent, stepparent, grandparent, other relative, or a foster parent, who has at least frequent contact with the subject. When possible both parents will participate in the assessment and treatment. Legal custody is always considered (e.g., divorced parents). Having all family members present at every session is not required. Many individual meetings with the subject or the parent are planned in both treatments.

Exclusion Criteria:

* Evidence of imminent risk of harm to self or others that cannot be safely treated on an outpatient basis
* Evidence of psychotic features [as reported on the Diagnostic Interview Schedule for Children; Voice Diagnostic Interview Schedule for Children (VDISC)]
* Evidence of suffering from severe cognitive impairment (e.g., mental retardation, severe developmental disorders) as evidenced by educational records, parental report and/or clinical impression).
* Subjects taking antidepressant medication for depression for less than 6 weeks prior to the screening.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Diamond, PhD, Principal Investigator — Drexel University; Roger Kobak, PhD, Principal Investigator — University of Delaware
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Beck AT, Brown GK, Steer RA. Psychometric characteristics of the Scale for Suicide Ideation with psychiatric outpatients. Behav Res Ther. 1997 Nov;35(11):1039-46. doi: 10.1016/s0005-7967(97)00073-9. PMID 9431735
- [Background] Restifo K, Bogels S. Family processes in the development of youth depression: translating the evidence to treatment. Clin Psychol Rev. 2009 Jun;29(4):294-316. doi: 10.1016/j.cpr.2009.02.005. Epub 2009 Mar 4. PMID 19356833
- [Background] Jensen PS. After TADS, can we measure up, catch up, and ante up? J Am Acad Child Adolesc Psychiatry. 2006 Dec;45(12):1456-60. doi: 10.1097/01.chi.0000237712.81378.9d. No abstract available. PMID 17135990
- [Background] Brent DA. Glad for what TADS adds, but many TADS grads still sad. J Am Acad Child Adolesc Psychiatry. 2006 Dec;45(12):1461-4. doi: 10.1097/01.chi.0000237708.28013.2a. No abstract available. PMID 17135991
- [Background] Beck, A., Steer, R. & Brown, G. (1996) The Beck Depression Inventory-Second Edition. San Antonio, TX: Psychological Corporation.
- [Background] Garber, J., Robinson, N.S., & Valentiner, D. (1997). The relation between parenting and adolescent depression: Self-worth as a mediator. Journal of Adolescent Research, 12, 12-33.
- [Background] Brent DA, Holder D, Kolko D, Birmaher B, Baugher M, Roth C, Iyengar S, Johnson BA. A clinical psychotherapy trial for adolescent depression comparing cognitive, family, and supportive therapy. Arch Gen Psychiatry. 1997 Sep;54(9):877-85. doi: 10.1001/archpsyc.1997.01830210125017. PMID 9294380
- [Background] Bloom BL. A factor analysis of self-report measures of family functioning. Fam Process. 1985 Jun;24(2):225-39. doi: 10.1111/j.1545-5300.1985.00225.x. PMID 4018243
- [Background] Reynolds, W., & Mazza, J. (1999). Assessment of suicidal ideation in inner-city children and young adolescents: Reliability and validity of the Suicidal Ideation Questionnaire-JR. School Psychology Review, 28, 17-30.
- [Derived] Abbott CH, Zisk A, Herres J, Diamond GS, Krauthamer Ewing S, Kobak R. Exploring the relations between interpersonal risk and adolescent suicidality during treatment. J Consult Clin Psychol. 2021 Jun;89(6):528-536. doi: 10.1037/ccp0000656. PMID 34264700
- [Derived] Ibrahim M, Levy S, Gallop B, Krauthamer Ewing S, Hogue A, Chou J, Diamond G. Therapist Adherence to Two Treatments for Adolescent Suicide Risk: Association to Outcomes and Role of Therapeutic Alliance. Fam Process. 2022 Mar;61(1):183-197. doi: 10.1111/famp.12660. Epub 2021 Apr 27. PMID 33904589
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] Zisk A, Abbott CH, Bounoua N, Diamond GS, Kobak R. Parent-teen communication predicts treatment benefit for depressed and suicidal adolescents. J Consult Clin Psychol. 2019 Dec;87(12):1137-1148. doi: 10.1037/ccp0000457. Epub 2019 Oct 24. PMID 31647277
- [Derived] Abbott CH, Zisk A, Bounoua N, Diamond GS, Kobak R. Predicting Patterns of Treatment Response and Outcome for Adolescents Who Are Suicidal and Depressed. J Am Acad Child Adolesc Psychiatry. 2019 Sep;58(9):897-906. doi: 10.1016/j.jaac.2018.12.013. Epub 2019 Mar 12. PMID 30877051
- [Derived] Diamond GS, Kobak RR, Krauthamer Ewing ES, Levy SA, Herres JL, Russon JM, Gallop RJ. A Randomized Controlled Trial: Attachment-Based Family and Nondirective Supportive Treatments for Youth Who Are Suicidal. J Am Acad Child Adolesc Psychiatry. 2019 Jul;58(7):721-731. doi: 10.1016/j.jaac.2018.10.006. Epub 2018 Oct 30. PMID 30768418
- [Derived] Bounoua N, Abbott C, Zisk A, Herres J, Diamond G, Kobak R. Emotion regulation and spillover of interpersonal stressors to postsession insight among depressed and suicidal adolescents. J Consult Clin Psychol. 2018 Jul;86(7):593-603. doi: 10.1037/ccp0000316. PMID 29939053

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Family-Enhanced Non-directive Supportive Therapy | Attachment-Based Family Therapy
Started | 63 | 66
Completed | 52 | 54
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Family-Enhanced Non-directive Supportive Therapy | Attachment-Based Family Therapy | Total
Number analyzed (Participants) | 63 | 66 | 129
Age, Customized [Count of Participants; unit: Participants]
  <=15 Years Old | 40 | 36 | 76
  >15 Years Old | 23 | 30 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 55 | 107
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 54 | 55 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 33 | 31 | 64
  White | 16 | 21 | 37
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 6 | 6 | 12
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 50 | 38 | 88
  Lesbian/Gay | 2 | 8 | 10
  Bisexual | 9 | 13 | 22
  Questioning | 2 | 7 | 9
Socioeconomic Status [Count of Participants; unit: Participants]
  Below Poverty Level | 19 | 21 | 40
  Above Poverty Level | 44 | 45 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change in the Intensity of Suicidal Ideation Between Intake and End of Treatment
Description: The Suicidal Ideation Questionnaire-JR is a 15-item self-report assessment. It is based on Reynolds' theoretical notion of suicidality forming a continuum ranging from thoughts of death, thoughts of wanting to be dead, general and specific suicidal plans, preparations for carrying out plans, and actual suicide attempts. The scale ranges from 0 to 90, with a score of 0 being representative of no suicidal ideation, and a score of 31 or greater indicating severe suicidal ideation.
Time Frame: 16 weeks (end of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family-Enhanced Non-directive Supportive Therapy | Attachment-Based Family Therapy
Number analyzed (Participants) | 52 | 54
units on a scale | -27.42 (2.52) | -31.55 (2.50)

2. Primary Outcome: Change in the Severity of Depression Symptoms Between Intake and End of Treatment
Description: Beck Depression Inventory-II. The second edition of the BDI is a widely-used, 21-item self-report instrument designed to assess the severity of depressive symptoms in adults and adolescents. The BDI-II has 21 items and takes approximately 5 minutes to complete. The scale ranges from 0 to 63, with a higher score being representative of a greater clinical magnitude of depression: a total score of 0-13 is considered minimal depression, 14-19 is mild depression, 20-28 is moderate depression, and 29-63 is severe depression.
Time Frame: 16 weeks (end of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family-Enhanced Non-directive Supportive Therapy | Attachment-Based Family Therapy
Number analyzed (Participants) | 52 | 54
units on a scale | -4.87 (0.50) | -5.40 (0.50)

3. Secondary Outcome: Change in the Evidence of Family Conflict Between Parent and Youth After Intervention Between Intake and End of Treatment
Description: The Self-Report of Family Functioning consists of 10 items selected from a number of well-known family assessment measures (Family Environment Scale, Family Concept Q-Sort, Family Adaptability and Cohesion Scale, and Family Assessment Measure). The scale ranges from 10 to 40, with a score of 10 being representative of no family conflict and a score of 40 being representative of the greatest magnitude of family conflict. Therefore, a decrease in score represents and decrease in self-reported family conflict.
Time Frame: 16 weeks (end of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family-Enhanced Non-directive Supportive Therapy | Attachment-Based Family Therapy
Number analyzed (Participants) | 53 | 55
units on a scale | -1.058 (2.95232) | -1.2538 (2.71817)

ADVERSE EVENTS:
Description: Given the definitions of expected outcomes, the following outcomes will be reported as SAEs if it is possible that they may be related to the completion of an assessment (e.g., participant becomes suicidal during or immediately following an assessment) or participation in treatment (e.g., participant becomes suicidal during or immediately following a treatment session): suicide attempt, death by suicide, psychiatric hospitalization.
Arm/Group | Family-Enhanced Non-directive Supportive Therapy | Attachment-Based Family Therapy
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/66
Other Adverse Events (participants affected / at risk) | 27/63 | 27/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family-Enhanced Non-directive Supportive Therapy (N=63) | Attachment-Based Family Therapy (N=66)
Suicide Attempt (Psychiatric disorders) | 3 (3) | 8 (10)
Non-suicidal self-injury (Psychiatric disorders) | 7 (9) | 7 (11)
Hospitalization (Psychiatric disorders) | 6 (6) | 2 (3)
Emergency Room Visit (Psychiatric disorders) | 1 (1) | 3 (3)
High level of suicidal ideation (Psychiatric disorders) | 11 (21) | 12 (23)
Abuse/Neglect (Psychiatric disorders) | 5 (9) | 3 (3)
Incarceration (Psychiatric disorders) | 0 (0) | 2 (2)
Other (Psychiatric disorders) | 7 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No